CLINICAL TRIAL: NCT02835027
Title: Treatment of Acute Lower Limb Ischaemia in Sweden 1994-2014
Status: Completed | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Martin Bjorck, Professor of Vascular Surgery, Uppsala University Hospital
Other Study IDs: Dnr2014/325
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Acute Ischemia of Lower Limb
Keywords: Acute limb ischaemia(ALI); Acute ischaemia of the lower extremity; Thrombosis; Emboli; Endovascular surgery; Surgery; Amputation free survival; Long time survival; Demographics
MeSH Terms: conditions — Thrombosis; Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 22 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Open versus endovascular surgery — Treatment for acute ischemia

SUMMARY:
Study of acute lower ischemia therapies based on data collected from the Swedish Vascular Surgery Registry between 1994 and 2014.

Primary endpoint is long term amputation-free survival and secondary end-points are 30 days and 1 year amputation-free survival as well as different revascularization techniques results and time trends.

DETAILED DESCRIPTION:
The prospective Swedish Vascular Registry (Swedvasc) started in 1987 and since 1994 it has included more than 95 percent of the vascular surgical procedures performed nationwide. The registry has received extensive high internal and external validation. Roughly 16000 open surgical and endovascular revascularisation procedures for acute limb ischemia have been performed during this period of time.

The fact that every Swedish citizen has a unique personal identification number makes it possible to obtain 100 percent accurate survival and amputation data. Survival data were obtained through crosschecking the personal identification number with the national population registry in June 2016.

This offers a unique opportunity to study a large population-based cohort of unselected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute limb ischemia
* Surgical procedure performed between 1 January 1994 and 31 December 2014 in Sweden and registered in the Swedvasc registry
* Infrainguinal occlusions

Exclusion Criteria:

* Acute limb ischemia secondary to trauma, bleedings, dissection or graft infections.
* Suprainguinal occlusions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The entire Swedish population, thus no sampling.
Sampling Method: Non-Probability Sample
Enrollment: 16287 (Actual)
Dates: Start 1994-01; Primary Completion 2014-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Amputation-free survival | 1-22 years
  Combined endpoint with death and amputation. Either the leg is amputated and/or the patient is dead or the patient is alive without major amputation.

SECONDARY OUTCOMES:
Amputation | 1-22 years
  Major amputation is defined as amputation above foot-level. Either the leg is amputated or not.
Survival | 1-22 years
  Either the patient is dead or alive
Complications 30 days after surgery | 30 days
  Bleeding, myocardial infarction, stroke, occlusion, compartment syndrome, etc

CONTACTS AND LOCATIONS:
Overall Officials: Martin Björck, Professor, Study Director — Uppsala University

IPD SHARING:
Plan to Share IPD: Undecided